CLINICAL TRIAL: NCT00151476
Title: A Registry-Based Observational Study Assessing Clinical Outcomes In Familial Adenomatous Polyposis In Patients Receiving Celecoxib (Celebrex(Registered), Onsenal(Registered)) Compared With Control Patients
Brief Title: Observational Familial Adenomatous Polyposis Registry Study In Patients Receiving Celecoxib Compared to Control Patients
Status: Terminated | Type: Observational
Why Stopped: See Detailed Description
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Other Study IDs: NQ4-00-02-012; A3191167
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Results first posted 2010-03-04 (Estimated); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Familial Adenomatous Polyposis (FAP)
Keywords: Familial adenomatous polyposis; celecoxib; IRA; IPAA
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Celecoxib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Celecoxib - Routine Medical Care: 800 mg total daily dosing
  Interventions: Drug: Celecoxib
- Control Group - Routine Medical Care: Observation of subjects treated with routine medical care
  Interventions: Other: Routine Medical Care

INTERVENTIONS:
Drug: Celecoxib — 800 mg total daily dosing
  Other Names: celebrex, SC-58635
  Groups: Celecoxib - Routine Medical Care
Other: Routine Medical Care
  Groups: Control Group - Routine Medical Care

SUMMARY:
This is a registry-based observational study assessing clinical outcomes in FAP patients receiving celecoxib compared with historical/concurrent registry patients who have not received celecoxib.

Both retrospective and prospective data will be utilized. No sampling methods apply.

DETAILED DESCRIPTION:
The study prematurely discontinued on April 11, 2008 due to slow enrollment. It should be noted that safety concerns have not been seen in this study and have not factored into this decision.

ELIGIBILITY:
Inclusion Criteria:

Celecoxib Treated Patients:

* Diagnosis of FAP based on the expression of the FAP phenotype.
* Celecoxib treatment prescribed outside of a clinical trial setting with expected duration of celecoxib treatment of at least six months.

Historical/Concurrent Control Patients:

* Diagnosis of FAP based on the expression of the FAP phenotype.
* Be greater than or equal to 12 years old at the time of study enrollment.
* Have an endoscopically assessable colonic, rectal, ileal pouch and/or gastroduodenal segment.
* For the group of post-surgical patients, IRA or IPAA performed from 1985 onward (in order to assure standardized surgical techniques and post-surgical management). Patients whose primary colorectal surgery was performed prior to 1985 will not be eligible to serve as historical controls.

Exclusion Criteria:

Celecoxib Treated Patients:

* Have received a pharmacological treatment (other than celecoxib) within the last 3 months for their FAP disease including treatment of any extracolonic manifestation of FAP.
* Have received a non-steroidal anti-inflammatory drug (NSAID) within the last 3 months, other than celecoxib, for any reason.

Historical/Concurrent Control Patients:

* Have pharmacological treatment recorded for their FAP disease at the defined index date.
* Have received a non-steroidal anti-inflammatory drug (NSAID) within the last 3 months for any reason.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with FAP
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2004-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Pfizer Investigational Site, Cleveland, Ohio, United States
- Pfizer Investigational Site, Toronto, Ontario, Canada
- Pfizer Investigational Site, Hvidovre, Copenhagen, Denmark
- Pfizer Investigational Site, Barcelona, Spain

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=NQ4-00-02-012&StudyName=Observational%20Familial%20Adenomatous%20Polyposis%20Registry%20Study%20In%20Patients%20Receiving%20Celecoxib

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study prematurely discontinued in May 2008 prior to reaching planned enrollment target; Last subject last visit November 2008.
Pre-assignment Details: Familial Adenomatous Polyposis (FAP) identified subjects=celecoxib-treated and matched control subjects eligible for inclusion in study identified from 4 registry sites; FAP analyzed=celecoxib-treated and matched control subjects eligible for matching and analysis in study. 1 subject excluded from analysis; took celecoxib without a prescription.
Groups:
- Matched Control: Observation of subjects not treated with celecoxib and followed according to routine medical practice; matched to matched celecoxib treated subjects. Routine medical practice: all patients regardless of treatment status are followed according to local standard of medical care by the respective physicians.
- All Celecoxib Treated: All celecoxib treated subjects (includes Matched Celecoxib Treated and Not Matched Celecoxib Treated subjects); treatment prescribed outside clinical trial setting per routine medical care. Routine medical care: celecoxib is prescribed in the usual manner in accordance with the terms of the marketing authorization and as prescribed in medical practice. The assignment of the patient to celecoxib is not decided in advance by the study protocol but falls within current practice. All patients regardless of treatment status are followed according to local standard of medical care by the respective physicians.
Period: FAP Identified Subjects
Arm/Group | Matched Control | All Celecoxib Treated
Started | 13 | 55
Completed | 13 | 54
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: FAP Analyzed Subjects
Arm/Group | Matched Control | All Celecoxib Treated
Started | 13 | 54
Completed | 13 | 51
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Other study participation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Matched Celecoxib Treated: Celecoxib treatment prescribed outside clinical trial setting per routine medical care; matched to control subjects. Routine medical care: celecoxib is prescribed in the usual manner in accordance with the terms of the marketing authorization and as prescribed in medical practice. The assignment of the patient to celecoxib is not decided in advance by the study protocol but falls within current practice. All patients regardless of treatment status are followed according to local standard of medical care by the respective physicians.
- Not Matched Celecoxib Treated: Celecoxib treatment prescribed outside clinical trial setting per routine medical care; not matched to control subjects. Routine medical care: celecoxib is prescribed in the usual manner in accordance with the terms of the marketing authorization and as prescribed in medical practice. The assignment of the patient to celecoxib is not decided in advance by the study protocol but falls within current practice. All patients regardless of treatment status are followed according to local standard of medical care by the respective physicians.
- Total: Total of all reporting groups
Arm/Group | Matched Celecoxib Treated | Matched Control | Not Matched Celecoxib Treated | Total
Number analyzed (Participants) | 13 | 13 | 41 | 67
Age, Customized [Number; unit: participants] — Age range groups at most recent FAP-related surgery (years). Prior to start of study follow-up = prior to baseline. Start of study follow-up: start of on-study celecoxib treatment period for celecoxib-treated subjects and index date for control subjects = baseline.
  participants
    <25 years | 4 | 5 | 18 | 27
    25 to 34 years | 5 | 4 | 5 | 14
    35 to 44 years | 3 | 2 | 8 | 13
    45 to 54 years | 1 (11.24) | 1 (9.00) | 3 | 5
    55 to 64 years | 0 | 0 | 1 | 1
    >64 years | 0 | 0 | 0 | 0
    Age not available (no surgery) | 0 | 1 | 6 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 21 | 29
  Male | 11 | 7 | 20 | 38

OUTCOME MEASURES:

1. Primary Outcome: Time From Ileorectal Anastomosis (IRA) to Time of First Excisional Polypectomy of a Rectal Polyp Post IRA
Description: Time(months): [date of first excisional polypectomy of rectal polyp post IRA minus date of prior IRA plus 1] divided by 30.44. Baseline = start of study follow-up: start of on-study celecoxib treatment period for celecoxib-treated subjects and comparable to index date for control subjects. Index date calculated as Matched Celecoxib-treated patients: number of days from most recent FAP-related surgery (IRA or IPAA) to start of study follow-up; add this number of days to matched control patient's most recent FAP-related surgery date=index date for Matched Control.
Time Frame: Up to 8 years prior to baseline
Population: All eligible subjects with IRA performed prior to start of study follow-up; first excisional polypectomy of rectal polyp post IRA. Polyp size unavailable for many subjects; not considered in analysis.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Matched Celecoxib Treated | Matched Control | Not Matched Celecoxib Treated | All Celecoxib Treated
Number analyzed (Participants) | 4 | 2 | 26 | 30
months | 86.4 (143.78) | 4.0 (3.25) | 78.4 (102.01) | 79.5 (105.44)
Statistical Analysis 1: Comparison: Matched Celecoxib Treated; Time to FAP-related surgical events (months); twenty-fifth (25th) percentile presented due to limited number of subjects. Index date based on most recent colon and or rectum adenomatous polyps evaluation, most recent duodenal adenomatous polyps evaluation, and most recent desmoids tumors evaluation for Matched Control, Not Matched Celecoxib, and All Celecoxib Treated, respectively. Only 13 matched pairs identified: p-values not computed in analysis of time-to-event endpoints; Test type: Superiority or Other; Kaplan-Meier Estimate of Time to Event = 14.49, 95% CI [3.48 to 301.64] — Kaplan-Meier Estimate of Time to Event (months)
Statistical Analysis 2: Comparison: Not Matched Celecoxib Treated; Time to FAP-related surgical events (months); 25th percentile; Test type: Superiority or Other; Kaplan-Meier Estimate of Time to Event = 5.06, 95% CI [3.48 to 11.76] — Kaplan-Meier Estimate of Time to Event (months)
Statistical Analysis 3: Comparison: All Celecoxib Treated; Time to FAP-related surgical events (months); 25th percentile; Test type: Superiority or Other; Kaplan-Meier Estimate of Time to Event = 5.52, 95% CI [3.48 to 14.49] — Kaplan-Meier Estimate of Time to Event (months)

2. Primary Outcome: Time From Start of Study Follow-up to the Time of First Excisional Polypectomy of a Rectal Polyp Post IRA
Description: Time(months): [date of first excisional polypectomy of rectal polyp post IRA minus date of start of study follow-up plus 1] divided by 30.44.
Time Frame: Baseline, Up to 60 months post-baseline
Population: All eligible subjects with IRA performed prior to start of study follow-up included, except left-censored subjects (had first excisional polypectomy of rectal polyp post IRA prior to start of study follow-up). No control group subjects (n=3) had a post-IRA polypectomy (no data).
Measure: Median (Full Range); unit: months
Arm/Group | Matched Celecoxib Treated | Matched Control | Not Matched Celecoxib Treated | All Celecoxib Treated
Number analyzed (Participants) | 1 | 0 | 5 | 6
months | 19.8 (17.14) [19.8 to 19.8] |  | 32.1 [0.0 to 44.1] | 25.9 [0.0 to 44.1]
Statistical Analysis 1: Comparison: Not Matched Celecoxib Treated; Time to FAP-related surgical events (months); 25th percentile; Test type: Superiority or Other; Kaplan-Meier Estimate of Time to Event = 5.98, 95% CI [0.00 to 33.77] — Kaplan-Meier Estimate of Time to Event (months)
Statistical Analysis 2: Comparison: All Celecoxib Treated; Time to FAP-related surgical events (months); 25th percentile; Test type: Superiority or Other; Kaplan-Meier Estimate of Time to Event = 19.81, 95% CI [0.00 to 33.77] — Kaplan-Meier Estimate of Time to Event (months)

3. Primary Outcome: Time From Ileopouch Anal Anastomosis (IPAA) to Time of First Excisional Polypectomy of a Rectal Polyp Post IPAA
Description: Time (months): [date of first excisional polypectomy of a rectal polyp post IPAA minus date of prior IPAA plus 1] divided by 30.44. Baseline = start of study follow-up: start of on-study celecoxib treatment period for celecoxib-treated subjects and comparable to index date for control subjects. Index date calculated as Matched Celecoxib-treated patients: number of days from most recent FAP-related surgery (IRA or IPAA) to start of study follow-up; add this number of days to matched control patient's most recent FAP-related surgery date=index date for Matched Control.
Time Frame: Up to 15 years prior to baseline
Population: All eligible subjects with IPAA performed prior to start of study follow-up included and with first excisional polypectomy of a rectal polyp post IPAA. No control group subjects (n=7) had a post-IPAA polypectomy (no data).
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Matched Celecoxib Treated | Matched Control | Not Matched Celecoxib Treated | All Celecoxib Treated
Number analyzed (Participants) | 3 | 0 | 0 | 3
months | 152.7 (42.10) |  |  | 152.7 (42.10)
Statistical Analysis 1: Comparison: Matched Celecoxib Treated; Time to FAP-related surgical events (months); 25th percentile. Index date based on most recent colon and or rectum adenomatous polyps evaluation, most recent duodenal adenomatous polyps evaluation, and most recent desmoids tumors evaluation for Matched Control, Not Matched Celecoxib, and All Celecoxib Treated, respectively; Test type: Superiority or Other; Kaplan-Meier Estimate of Time to Event = 137.34, 95% CI [104.73 to 183.48] — Kaplan-Meier Estimate of Time to Event (months)
Statistical Analysis 2: Comparison: All Celecoxib Treated; Time to FAP-related surgical events (months); 25th percentile; Test type: Superiority or Other; Kaplan-Meier Estimate of Time to Event = 169.94, 95% CI [104.73 to 183.48] — Kaplan-Meier Estimate of Time to Event (months)

4. Primary Outcome: Time From Start of Study Follow-up to Time of First Excisional Polypectomy of a Rectal Polyp Post IPAA
Description: Time (months): [date of first excisional polypectomy of rectal polyp post IPAA minus date of start of study follow-up plus 1] divided by 30.44.
Time Frame: Baseline, Up to 60 months post-baseline
Population: All eligible subjects with IPAA performed prior to start of study follow-up included, except left-censored subjects (had first excisional polypectomy post IPAA prior to start of study follow-up). No control group subjects (n=7) had a post-IPAA polypectomy (no data).
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Matched Celecoxib Treated | Matched Control | Not Matched Celecoxib Treated | All Celecoxib Treated
Number analyzed (Participants) | 3 | 0 | 0 | 3
months | 20.3 (15.72) |  |  | 20.3 (15.72)
Statistical Analysis 1: Comparison: Matched Celecoxib Treated; Time to FAP-related surgical events (months); 25th percentile; Test type: Superiority or Other; Kaplan-Meier Estimate of Time to Event = 11.28, 95% CI [9.07 to 38.24] — Kaplan-Meier Estimate of Time to Event (months)

5. Secondary Outcome: Time From Most Recent Prior FAP-related Surgical Event or Onset of FAP Phenotype to Time of First Excisional or Ablational Event for Rectal, Colonic, Pouch, or Duodenal Adenomas (Duodenal Adenomatous Polyps)
Description: Time (months): [date of first excisional or ablational event for colonic, pouch, or duodenal adenomas occuring after date of most recent prior FAP-related surgical event or date of FAP diagnosis minus date of most recent prior FAP-related surgical event or date of FAP diagnosis plus 1] divided by 30.44.
Time Frame: Up to 15 years prior to baseline
Population: All eligible subjects; first excisional or ablational event for rectal adenomas that does not qualify for primary efficacy endpoint; after most recent FAP-related surgical event prior to start of study follow-up or onset of FAP phenotype for subjects with no prior FAP-related surgery.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Matched Celecoxib Treated | Matched Control | Not Matched Celecoxib Treated | All Celecoxib Treated
Number analyzed (Participants) | 8 | 8 | 33 | 41
months | 25.7 (18.71) | 47.7 (42.32) | 89.9 (89.34) | 77.4 (84.32)
Statistical Analysis 1: Comparison: Matched Celecoxib Treated; Time to FAP-related surgical events (months); 25th percentile; Test type: Superiority or Other; Kaplan-Meier Estimate of Time to Event = 20.63, 95% CI [8.05 to 48.03] — Kaplan-Meier Estimate of Time to Event (months)
Statistical Analysis 2: Comparison: Matched Control; Time to FAP-related surgical events (months); 25th percentile; Test type: Superiority or Other; Kaplan-Meier Estimate of Time to Event = 40.21, 95% CI [8.31 to 105.68] — Kaplan-Meier Estimate of Time to Event (months)
Statistical Analysis 3: Comparison: Not Matched Celecoxib Treated; Time to FAP-related surgical events (months); 25th percentile; Test type: Superiority or Other; Kaplan-Meier Estimate of Time to Event = 19.81, 95% CI [16.03 to 56.34] — Kaplan-Meier Estimate of Time to Event (months)
Statistical Analysis 4: Comparison: All Celecoxib Treated; Time to FAP-related surgical events (months); 25th percentile; Test type: Superiority or Other; Kaplan-Meier Estimate of Time to Event = 20.22, 95% CI [12.35 to 40.31] — Kaplan-Meier Estimate of Time to Event (months)

6. Secondary Outcome: Time From Start of Study Follow-up to Time of First Excisional or Ablational Event for Rectal, Colonic, Pouch, or Duodenal Adenomas
Description: Time (months): [date of first excisional or ablational event for colonic, pouch, or duodenal adenomas, occurring after date of most recent prior FAP-related surgical event, or date of FAP diagnosis minus date of start of study follow-up plus 1] divided by 30.44.
Time Frame: Baseline, Up to 60 months post-baseline
Population: All eligible subjects included, except left censored subjects (had any excisional or ablational event for rectal, colonic, pouch, or duodenal adenomas between date of most recent FAP-related surgical event performed prior to the start of study follow-up, or onset of FAP phenotype [with no prior FAP-related surgery], and start of study follow-up).
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Matched Celecoxib Treated | Matched Control | Not Matched Celecoxib Treated | All Celecoxib Treated
Number analyzed (Participants) | 2 | 3 | 3 | 5
months | 0.0 (0.0) | 41.7 (21.73) | 21.4 (22.39) | 12.9 (19.71)

7. Secondary Outcome: Time From Most Recent Prior FAP-related Surgical Event or Onset of FAP Phenotype to Time of First FAP-related Adverse Event
Description: Time (months): [date of first FAP-related adverse event, occurring after the date of most recent prior FAP-related surgery, or date of FAP diagnosis minus date of most recent prior FAP-related surgery, or date of FAP diagnosis plus 1] divided by 30.44. FAP-related adverse event defined as any FAP related cancers, desmoid tumors requiring procedural intervention, hospitalizations or procedural interventions, or death related to FAP (i.e., as a consequence of FAP, FAP complications, or a procedure or drug used to treat FAP-related medical problems).
Time Frame: Up to 15 years prior to baseline
Population: All eligible subjects; first FAP-related adverse event (FAP-related cancers, desmoid tumors requiring procedural intervention, hospitalizations, procedural interventions, or death related to FAP) after subject's most recent FAP-related surgical event performed prior to start of study follow-up, onset of FAP phenotype (no prior FAP-related surgery).
Measure: Median (Full Range); unit: months
Arm/Group | Matched Celecoxib Treated | Matched Control | Not Matched Celecoxib Treated | All Celecoxib Treated
Number analyzed (Participants) | 5 | 6 | 30 | 35
months | 3.0 (123.17) [0.2 to 167.0] | 3.4 (48.34) [2.5 to 123.8] | 61.4 [1.1 to 362.9] | 56.3 [0.2 to 362.9]
Statistical Analysis 1: Comparison: Not Matched Celecoxib Treated; Time to FAP-related events (months); 25th percentile; Test type: Superiority or Other; Kaplan-Meier Estimate of Time to Event = 21.22, 95% CI [4.07 to 64.16] — Kaplan-Meier Estimate of Time to Event (months)
Statistical Analysis 2: Comparison: All Celecoxib Treated; Time to FAP-related events (months); 25th percentile; Test type: Superiority or Other; Kaplan-Meier Estimate of Time to Event = 19.81, 95% CI [3.68 to 64.16] — Kaplan-Meier Estimate of Time to Event (months)

8. Secondary Outcome: Time From Start of Study Follow-up to Time of First FAP-related Adverse Event
Description: Time (months): [date of first FAP-related adverse event, occurring after the date of the most recent prior FAP-related surgery, or date of FAP diagnosis minus date of start of study follow-up plus 1] divided by 30.44. FAP-related adverse event defined as any FAP related cancers, desmoid tumors requiring procedural intervention, hospitalizations or procedural interventions, or death related to FAP (i.e., as a consequence of FAP, FAP complications, or a procedure or drug used to treat FAP-related medical problems).
Time Frame: Baseline, Up to 60 months post-baseline
Population: All eligible subjects included, except left-censored subjects (had any FAP-related adverse event between the date of most recent FAP-related surgical event performed prior to start of study follow-up, or onset of FAP phenotype (no prior FAP-related surgery), and start of study follow-up.
Measure: Median (Full Range); unit: months
Arm/Group | Matched Celecoxib Treated | Matched Control | Not Matched Celecoxib Treated | All Celecoxib Treated
Number analyzed (Participants) | 1 | 1 | 7 | 8
months | 37.9 [37.9 to 37.9] | 75.7 [75.7 to 75.7] | 9.7 [0.8 to 37.7] | 14.3 [0.8 to 37.9]

9. Secondary Outcome: Time From Post IRA to Time of Conversion From IRA to IPAA
Description: Time (months): [date of IPAA minus date of prior IRA plus 1] divided by 30.44.
Time Frame: Up to 15 years prior to baseline
Population: All eligible subjects with IRA performed prior to start of study follow-up; data censored (n=5) for control group subjects (no data).
Measure: Median (Full Range); unit: months
Arm/Group | Matched Celecoxib Treated | Matched Control | Not Matched Celecoxib Treated | All Celecoxib Treated
Number analyzed (Participants) | 1 | 0 | 9 | 10
months | 301.6 [301.6 to 301.6] |  | 129.7 [8.0 to 362.9] | 175.8 [8.0 to 362.9]

10. Secondary Outcome: Time From Start of Study Follow-up to Time of Conversion From IRA to IPAA
Description: Time (months): [date of IPAA minus date of start of study follow-up plus 1] divided by 30.44.
Time Frame: Baseline, Up to 60 months post-baseline
Population: All eligible subjects with IRA performed prior to start of study follow-up included, except left-censored subjects (had IPAA prior to start of study follow-up); data censored (n=5) for control group subjects (no data).
Measure: Median (Full Range); unit: months
Arm/Group | Matched Celecoxib Treated | Matched Control | Not Matched Celecoxib Treated | All Celecoxib Treated
Number analyzed (Participants) | 0 | 0 | 2 | 2
months |  |  | 4.8 [0.0 to 9.7] | 4.8 [0.0 to 9.7]

11. Post Hoc Outcome: Duodenal Adenoma Burden as Measured by Polyp Counts
Description: Number of subjects with polyp burden as assessed in most recent prior polyps evaluation: attenuated: <100 polyps, mild: between 100 to 1000 polyps, severe: >1000 polyps. EOS: endoscopic examination closest to end of on-study celecoxib or index period (within 6 months of end of celecoxib or index period and prior to intake of any exclusionary medications after baseline). Post-hoc analysis of duodenal polyp burden in terms of severity categories and based on polyp numbers; Spigelman Stage not completed as staging data largely missing (see: Duodenal adenoma burden as measured by Spigelman Stage)
Time Frame: Baseline, 6 to 14 months post-baseline, End of study (EOS)
Population: All subjects; Spigelman Stage not completed as staging data largely missing; duodenal polyp burden analyzed in terms of severity categories and based on polyp numbers.
Measure: Number; unit: participants
Arm/Group | Matched Celecoxib Treated | Matched Control | Not Matched Celecoxib Treated | All Celecoxib Treated
Number analyzed (Participants) | 13 | 13 | 41 | 54
participants
  Baseline attenuated | 5 | 1 | 18 | 23
  Baseline mild | 0 | 0 | 0 | 0
  Baseline severe | 0 | 0 | 0 | 0
  Baseline unknown | 3 | 2 | 10 | 13
  Baseline no polyps | 1 | 5 | 5 | 6
  Baseline not assessed | 4 | 5 | 8 | 12
  Post-baseline attenuated | 1 | 3 | 12 | 13
  Post-baseline mild | 0 | 0 | 0 | 0
  Post-baseline severe | 0 | 0 | 0 | 0
  Post-baseline unknown | 3 | 0 | 0 | 3
  Post-baseline no polyps | 1 | 3 | 0 | 1
  Post-baseline not assessed | 8 | 7 | 29 | 37
  EOS attenuated | 2 | 2 | 17 | 19
  EOS mild | 0 | 0 | 0 | 0
  EOS severe | 0 | 0 | 0 | 0
  EOS unknown | 1 | 0 | 2 | 3
  EOS no polyps | 1 | 1 | 2 | 3
  EOS not assessed | 9 | 10 | 20 | 29

12. Secondary Outcome: Duodenal Adenoma Burden as Measured by Spigelman Stage
Description: Number of subjects with polyp burden as assessed in most recent prior polyps evaluation: Spigelman stage provides index of disease severity based on number of polyps, polyp size, histology, and dysplasia; range is Stage 0 (none) to Stage IV (severe). EOS: endoscopic examination closest to end of on-study celecoxib or index period (within 6 months of end of celecoxib or index period and prior to intake of any exclusionary medications after baseline). Spigelman Stage not completed as staging data largely missing; see measure: Duodenal adenoma burden as measured by polyp counts.
Time Frame: Baseline, 6 to 14 months post-baseline, End of study (EOS)
Population: All subjects; Spigelman Stage not completed as staging data largely missing.
Arm/Group | Matched Celecoxib Treated | Matched Control | Not Matched Celecoxib Treated | All Celecoxib Treated
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Rectal or Pouch Adenoma Burden Based on Polyp Counts
Description: Number of subjects with polyp burden as assessed in most recent prior polyps evaluation: attenuated: <100 polyps, mild: between 100 to 1000 polyps, severe: >1000 polyps. EOS: endoscopic examination closest to end of on-study celecoxib or index period (within 6 months of end of celecoxib or index period and prior to intake of any exclusionary medications after baseline).
Time Frame: Baseline, 6 to 14 months post-baseline, EOS
Population: All subjects; duodenal polyp burden analyzed in terms of severity categories and based on polyp numbers.
Measure: Number; unit: particpants
Arm/Group | Matched Celecoxib Treated | Matched Control | Not Matched Celecoxib Treated | All Celecoxib Treated
Number analyzed (Participants) | 13 | 13 | 41 | 54
particpants
  Baseline attenuated | 9 | 4 | 18 | 27
  Baseline mild | 2 | 2 | 2 | 4
  Baseline severe | 0 | 0 | 0 | 0
  Baseline unknown | 1 | 0 | 12 | 13
  Baseline no polyps | 1 | 6 | 4 | 5
  Baseline not assessed | 0 | 1 | 5 | 5
  Post-baseline attenuated | 6 | 3 | 10 | 16
  Post-baseline mild | 0 | 0 | 1 | 1
  Post-baseline severe | 0 | 0 | 0 | 0
  Post-baseline unknown | 0 | 0 | 0 | 0
  Post-baseline no polyps | 4 | 5 | 1 | 5
  Post-baseline not assessed | 3 | 5 | 29 | 32
  EOS attenuated | 8 | 2 | 12 | 20
  EOS mild | 0 | 0 | 0 | 0
  EOS severe | 0 | 0 | 0 | 0
  EOS unknown | 3 | 0 | 1 | 4
  EOS no polyps | 2 | 6 | 2 | 4
  EOS not assessed | 0 | 5 | 26 | 26

ADVERSE EVENTS:
Time Frame: Up to 15 years prior to baseline; up to 5 years post-baseline. No safety information actively searched for among celecoxib-treated subjects for retrospectively collected data (medical records); if serious adverse event (SAE) found, it was reported as SAE.
Description: All SAEs, expected and unexpected, occurring while subject was receiving celecoxib during his/her prospective (on-study) participation in the study, regardless of the apparent relationship to the drug, were collected and reported to the sponsor. Not applicable to Matched Control subjects n=13; SAEs not collected if no celecoxib treatment received.
Arm/Group | All Celecoxib Treated
Serious Adverse Events (participants affected / at risk) | 5/54
Other Adverse Events (participants affected / at risk) | 0/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Celecoxib Treated (N=54)
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Duodenal perforation (Gastrointestinal disorders) | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Study prematurely discontinued May 2008 prior to reaching enrollment target; due to limited number of matched pairs, results do not provide sufficient data to evaluate effectiveness of celecoxib. Last subject last visit was November 2008.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.